CLINICAL TRIAL: NCT01263288
Title: Effect of Vitamin D Supplementation on Muscular Strength, Musculoskeletal Pain and Headache in Immigrants Living in Norway. Randomized, Double Blinded, Placebo Controlled Study
Brief Title: Effect of Vitamin D Supplementation on Muscular Strength, Musculoskeletal Pain and Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Per Lagerlov (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor-Investigator, Per Lagerlov, Associate Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2010-1982
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Vitamin Deficiency
MeSH Terms: conditions — Avitaminosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D3 (cholecalciferol) 400 IU (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol
- Vitamin D3 (cholecalciferol) 1000 IU (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Vitamin D3 tablet 400 IU. Once daily by mouth for 4 months
  Other Names: NN007
  Arms: Vitamin D3 (cholecalciferol) 400 IU
Dietary Supplement: cholecalciferol — Vitamin D3 tablet 1000 IU. Once daily by mouth for 4 months
  Other Names: NN008
  Arms: Vitamin D3 (cholecalciferol) 1000 IU
Dietary Supplement: Placebo — Microcrystalline cellulose tablet p.o.daily. (Same color, shape and size as vitamin D tablet)
  Other Names: NN009
  Arms: Placebo

SUMMARY:
The primary aim of the present trial is to study the effect of daily vitamin D supplementation on muscular power and force among non-western immigrants living in Oslo, Norway, and secondarily to study the effect of musculoskeletal pain and headache.

The investigators have also prespecified a number of additional research questions about anemia, metabolism and bone turnover, inflammation, diabetes, lipids, itching and kidney function, which because of multiple comparisons should be interpreted with caution unless the statistical evidence for an effect is very strong.

DETAILED DESCRIPTION:
Vitamin D deficiency is a widespread public health problem among immigrants from non-Western countries in Norway. As a background for preventive strategies it is important to have best possible knowledge about health consequences of poor vitamin D status, and in this respect much is lacking.

The investigators will aim to study the effect of vitamin D supplementation on muscular strength , musculoskeletal pain and headache among non-western immigrants in Norway with background from Middle East, Africa and South Asia. In addition the intervention gives us the opportunity to study the effect of vitamin D on indicators of other important health issues including anemia, diabetes , lipids, inflammation, metabolism and bone health. The study will also contribute with insight on how to achieve a high compliance. This is of interest in a broader context as poor compliance has been experienced as a problem in primary health care among immigrants with poor vitamin D status.

The study is a randomized, double blinded, placebo-controlled trial which compares two doses of vitamin D supplements, 400 IU and 1000 IU, with placebo and the tablets will be taken daily in a period of 4 months. Three muscle strength tests will be used, and they will be performed before and after the intervention: Counter movement jumps, Chair rising and Handgrip. Level and location of musculoskeletal pain and headache will be recorded at baseline and at end of the study.

A blood sample will be collected from the study subjects at baseline and after 4 months. The level of vitamin D and markers of anemia, metabolism and bone turnover, inflammation, diabetes, lipids and kidney function will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 - 50 years old
* Immigrants with background from Middle East, Africa and South Asia.

Exclusion Criteria:

* Daily use of vitamin D supplementation and frequently use of artificial UV light exposure.
* Pregnancy
* Malabsorptive disorders
* Fracture in the leg /arm within the preceding 6 months. Known osteoporosis
* Tuberculosis, sarcoidosis, cancer, kidney dysfunction, liver dysfunction and history of kidney stone.
* Regular use of medication that interfere with vitamin D/bone metabolism, such as glucocorticoids, diuretics, lithium, antiepileptics, bisphosphonates,
* Regular use of strong pain killers.
* Medication for diabetes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Muscular strength: jump height | 4 months

SECONDARY OUTCOMES:
Musculoskeletal pain, headache, muscular strength; chair rising and handgrip | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Lagerlov, MD, PhD, Study Chair — University of Oslo; Haakon E Meyer, Professor, Study Chair — University of Oslo
Locations (1):
- University of Oslo, Institute of Health and Society, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Knutsen KV, Brekke M, Gjelstad S, Lagerlov P. Vitamin D status in patients with musculoskeletal pain, fatigue and headache: a cross-sectional descriptive study in a multi-ethnic general practice in Norway. Scand J Prim Health Care. 2010 Sep;28(3):166-71. doi: 10.3109/02813432.2010.505407. PMID 20642395
- [Derived] Madar AA, Knutsen KV, Stene LC, Brekke M, Lagerlov P, Meyer HE, Macdonald HM. Effect of vitamin D3-supplementation on bone markers (serum P1NP and CTX): A randomized, double blinded, placebo controlled trial among healthy immigrants living in Norway. Bone Rep. 2015 May 21;2:82-88. doi: 10.1016/j.bonr.2015.05.004. eCollection 2015 Jun. PMID 28377958
- [Derived] Madar AA, Knutsen KV, Stene LC, Brekke M, Meyer HE, Lagerlov P. Effect of vitamin D3 supplementation on glycated hemoglobin (HbA1c), fructosamine, serum lipids, and body mass index: a randomized, double-blinded, placebo-controlled trial among healthy immigrants living in Norway. BMJ Open Diabetes Res Care. 2014 Oct 13;2(1):e000026. doi: 10.1136/bmjdrc-2014-000026. eCollection 2014. PMID 25452867
- [Derived] Knutsen KV, Madar AA, Lagerlov P, Brekke M, Raastad T, Stene LC, Meyer HE. Does vitamin D improve muscle strength in adults? A randomized, double-blind, placebo-controlled trial among ethnic minorities in Norway. J Clin Endocrinol Metab. 2014 Jan;99(1):194-202. doi: 10.1210/jc.2013-2647. Epub 2013 Dec 20. PMID 24248184